CLINICAL TRIAL: NCT00204321
Title: Influence of Sirolimus and MMF on Vascular Function and Markers of Cellular Function in Renal Transplant Recipients - Positive Effects of Calcineurin-free Immunosuppression
Brief Title: Influence of Sirolimus and MMF on Vascular Function and Markers of Cellular Function in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Prof. Dr. Hausberg, UKM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hausberg_Lang-Sir/MMF; EKF Hausberg Lang
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Renal Transplantation
Keywords: rejection; vesselwall function; endothelial cell function; monocytes
MeSH Terms: conditions — Rejection, Psychology | interventions — Sirolimus; Pharmaceutical Preparations; Mycophenolic Acid

INTERVENTIONS:
Drug: sirolimus (drug), mmf (drug)

SUMMARY:
Chronic transplant nephropathy and cardiovascular death are the main reasons for loss of transplanted organs after kidney transplantation.

Vascular changes, induced by hypertension and/or immunological processes, determine long time transplant survival.

It will be tested whether the withdrawal of calcineurininhibitors will improve the vessel wall function in renal transplant patients. It is supposed that this immunosuppressive regimen reduces the activation of endothelial cells with important impact on arteriosclerosis and therefore on patient and transplant survival.

DETAILED DESCRIPTION:
Cardiovascular complications and chronic rejection are chief causes of transplant loss[1,2]. After renal transplantation patients are still characterized by their pre-existing arteriosclerotic changes [3]. Endothelial dysfunction and disturbed distensibility of great arteries are independent predictors of cardiovascular morbidity [4,5]. Additionally the activation of sympathetic nervous system leads to dysfunction of vessel wall[6,7]. There are important therapeutic options in improvement of endothelial function [8].

In addition monocytes of the recipient will contribute to vessel wall changes. [9-11]. Aim of therapy - especially of immunosuppressive therapy- have to prevent these fatal vessel wall changes.

Therefore in this study the following topics will be addressed.

1. Discontinuing of calcineurininhibitors will lead to improvement of vessel wall function 2. Sirolimus and Mycophenolat Mofetil affect vessel wall properties in a different way.

3. There are risk factors, e.g. activity of sympathetic nervous system, which may determine the efficacy of discontinuing the calcineurininhibitor concerning the vessel wall function.

4. Calcineurininhibitorfree immunosuppression reduces the activity of endothelial cells.

5. Survival of monocytes and release of procoagulatory activity will be changed by the immunosuppressive regimen.

1. Rostand SG, Brunzell JD, Cannon RO, Victor RG. Cardiovascular complications in renal failure. J Am Soc Nephrol. 1991; 2: 1053-1062
2. London GM, Druecke TB. Atherosclerosis and arteriosclerosis in chronic renal failure. Kidney Int 1997; 51(6):1678-1695.
3. Hausberg, M., K. Kisters, M. Kosch, K. H. Rahn, and M. Barenbrock. Flow-mediated vasodilation and distensibility of the brachial artery in renal allograft recipients. Kidney Int. 55: 1104-1110, 1999.
4. Barenbrock M, Kosch M, Jöster E, Kisters K, Rahn KH, Hausberg M: Reduced arterial distensibility is a predictor of cardiovascular disease in patients after renal transplantation. Journal of Hypertension 2002, 20:79-84.
5. London GM, Pannier B, Agharazii M, Guerin AP, Verbeke FHM, Marchais SY. Forearm reactive hyperemia and mortality in end-stage-disease. Kidney Int 2004, 65:700-704.
6. Converse RL, Jacobsen TN, Toto RD, Jost CMT, Cosentino F, Fouad-Tarazi F, Victor RG. Sympathetic overactivity in patients with chronic renal failure. N Engl J Med 1992; 327:1912-1918.
7. Hausberg M, Kosch M, Harmelink P, Barenbrock M, Hohage H, Kisters K, Dietl KH, Rahn KH. Sympathetic nerve activity in end-stage renal disease. Circulation. 2002, 106:1974-9.
8. Kosch M, Barenbrock M, Kisters K, Rahn KH, Hausberg M. Relationship between muscle sympathetic nerve activity and large artery mechanical vessel wall properties in renal transplant patients. J Hypertens. 2002, 20:501-8.
9. Österud, A., Björklid E. Role of monocytes in atherogenesis. Physiological reviews, 2003, 83: 1069-1112.
10. Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26.
11. Lessner SM, Prado HL, Waller EK, Galis ZS. Atherosclerotic lesions grow through recruitment and proliferation of circulating monocytes in a murine model. Am J Pathol. 2002 Jun;160(6):2145-55.

ELIGIBILITY:
Inclusion Criteria:

renal transplantation stable function

Exclusion Criteria:

acute rejection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
distensibility
sympathetic nervous system activity
endothelial cell marker expression

SECONDARY OUTCOMES:
monocyte survival

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hausberg, MD, Principal Investigator — UKM - Medical Department D
Locations (1):
- UKM, Münster, North Rhine-Westphalia, Germany